CLINICAL TRIAL: NCT06017479
Title: Effectiveness of Single Dose Fosfomycin and Single Dose Levofloxacin as Pre-urodynamic Antibiotic Prophylaxis for Urinary Tract Infection Prevention in Post-Urodynamic Examination
Brief Title: Effectiveness of Single Dose Fosfomycin and Single Dose Levofloxacin as Pre-urodynamic Antibiotic for UTI Prevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Harrina Erlianti Rahadjo, Sp.U(K), PhD, Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-11-1343
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Urological System Complication of Procedure; Urinary Tract Infections
Keywords: urodynamic; urinary tract infections; fosfomycin; levofloxacin
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with a single-blinded randomized clinical trial design to compare the proportion of UTIs in a group of patients receiving fosfomycin 3 grams and patients receiving levofloxacin 500 miligrams single dose one hour before urodynamic examination. To determine the sample treatment group, blocked randomization technique is used in this study.
Who Masked: Outcomes Assessor
Masking Description: This study uses a single-blinded design because the outcome assessed in this study is urinalysis which is the objective outcome. The urinalysis evaluator is blinded to the drug regimen obtained by the research subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-urodynamic Fosfomycin (Experimental): Fosfomycin 3 g single dosage 1 hour before the urodynamic examination
  Interventions: Drug: Fosfomycin 3000 MG
- Pre-urodynamic Levofloxacin (Experimental): Levofloxacin 500 miligrams single dosage 1 hour before the urodynamic examination
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Fosfomycin 3000 MG — Fosfomycin 3 g single dosage 1 hour before the urodynamic examination
  Other Names: Monuril
  Arms: Pre-urodynamic Fosfomycin
Drug: Levofloxacin 500mg — Levofloxacin 500 mg single dosage 1 hour before the urodynamic examination
  Other Names: Levaquin
  Arms: Pre-urodynamic Levofloxacin

SUMMARY:
The goal of this clinical trial is to compare the use of single dose fosfomycin and single dose levofloxacin as pre-urodynamic antibiotic prophylaxis for urinary tract infection prevention post-urodynamic in patients with lower urinary tract symptoms. The main question[s] it aims to answer are:

* What is the difference between the effectiveness of administering a single dose of fosfomycin and levofloxacin prior to the procedure in terms of the incidence rate of urinary tract infection (UTI) post-urodynamic examination?
* What is the incidence rate of UTI in the administration of single-dose fosfomycin and levofloxacin prior to the procedure on the incidence rate of UTI post-urodynamic examination? Participants fulfilling the inclusion criteria will be taken their history and vital signs and consume either fosfomycin or levofloxacin based on the randomisation prior to urodynamic procedure. Afterwards, participants will undergo urine analysis 4 days post urodynamic to evaluate if there's any urinary tract infection. If there is any bacteria present, the sample will be cultured to identify bacteria found in the urine.

DETAILED DESCRIPTION:
This study employs a single-blinded randomized clinical trial design to compare the proportion of UTI post-urodynamic examination between the group receiving single-dose levofloxacin pre-urodynamic examination and the group receiving levofloxacin post-urodynamic examination for three days. The target population consists of patients undergoing urodynamic examination at Dr. Cipto Mangunkusumo National Referral Hospital, Persahabatan National Hospital, and Siloam Asri Hospital. The total sample size required for this study is 126 patients. On the fourth day post-urodynamic examination, urinalysis and urine culture are performed to determine the diagnosis of UTI. To analyze the association between UTI and therapy groups, a chi-square test is used. Results are considered statistically significant if p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients > 18 years who have indications for urodynamics
* Willing to participate in research

Exclusion Criteria:

* Allergy to levofloxacin
* Allergy to fosfomycin
* History of taking antibiotics in 1 month
* Pregnant
* Uncontrolled DM
* Use of urinary catheter
* Having a UTI before urodynamics, based on clinical symptoms and urine examination results
* Refuse to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harrina E Rahardjo, Professor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
These are the study protocol used in this study
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Rahardjo HE, Tirtayasa PM, Afriansyah A, Parikesit D, Akbar MI. The Effectiveness of a Three Day Course Antibiotic Post-urodynamic Study in Preventing Lower Urinary Tract Infection. Acta Med Indones. 2016 Apr;48(2):84-90. PMID 27550876
- [Background] Chu CM, Lowder JL. Diagnosis and treatment of urinary tract infections across age groups. Am J Obstet Gynecol. 2018 Jul;219(1):40-51. doi: 10.1016/j.ajog.2017.12.231. Epub 2018 Jan 2. PMID 29305250
- [Background] Fajfr M, Balik M, Cermakova E, Bostik P. Effective Treatment for Uncomplicated Urinary Tract Infections with Oral Fosfomycin, Single Center Four Year Retrospective Study. Antibiotics (Basel). 2020 Aug 13;9(8):511. doi: 10.3390/antibiotics9080511. PMID 32823650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected using consecutive sampling until the required number of subjects was reached. The primary data source is from patients with indications for urodynamic examination at Dr. Cipto Mangunkusumo, Siloam Asri, and Persahabatan Hospitals, starting December 30, 2022.
Pre-assignment Details: The inclusion criteria were any above 18-year-old who underwent UDS & were willing to participate in this study. Patients who had at least one of these exclusion criteria were excluded: allergy to levofloxacin, history of antibiotics consumption in 1 month prior to the study, pregnancy, uncontrolled and untreated diabetes mellitus, use of urinary catheter, UTI proved through urinalysis prior to the study, and refusal to participate.
Period: Overall Study
Arm/Group | Pre-urodynamic Fosfomycin | Pre-urodynamic Levofloxacin
Started | 63 | 63
Completed | 63 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Besides the required samples are 126 samples to complete the study. There are 59 samples that didn't meet the inclusion criteria of the study, which are because of there are 8 samples who refuse to participate, 14 samples that are under 18 years old, 7 samples that have history of antibiotics consumption in 1 month prior to the study, 19 samples that are UTI proved through urinalysis, 11 samples that use of urinary catheter prior to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-urodynamic Fosfomycin | Pre-urodynamic Levofloxacin | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.99 (19.08) | 42 (17.17) | 52.2 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 36 | 39 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 63 | 63 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Main Outcome Measure Was the Incidence of Urinary Tract Infection (UTI) Post-urodynamic Study (UDS), Diagnosed Through Urinalysis Indicating Leukocyturia, Positive Bacteria, Nitrite, and/or Leukocyte Esterase, Along With Clinical Symptoms.
Description: Urinary tract infections (UTIs) were diagnosed using a combination of urinalysis and clinical symptoms. A positive result was determined by leukocyturia (more than five white blood cells per field of vision), presence of bacteria, nitrite, and/or leukocyte esterase. Patients diagnosed with UTI underwent urine cultures to identify bacterial presence and determine the specific pathogen. The study used descriptive statistics to compare UTI incidences between the two treatment groups (levofloxacin vs. fosfomycin), and statistical significance was assessed using chi-square analysis with a p-value of <0.05.
Time Frame: 4 days post-urodynamic procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-urodynamic Fosfomycin | Pre-urodynamic Levofloxacin
Number analyzed (Participants) | 63 | 63
Participants
  Diagnosed UTI | 12 | 14
  Symptomatic UTIs | 7 | 6
  Non UTIs | 44 | 43
Statistical Analysis 1: Comparison: Pre-urodynamic Fosfomycin vs Pre-urodynamic Levofloxacin; This randomized controlled trial compared the incidence of UTI between two groups: patients receiving a single dose of 500 mg levofloxacin and patients receiving a single dose of 3 g fosfomycin one hour before a urodynamic study. The null hypothesis is that there is no significant difference in UTI incidence between the two groups. The power calculation was based on a sample size of 126 patients; Test type: Other — "Chi-square test" as the study used chi-square analysis to compare the incidence of UTIs between the groups (p = 0.660) For this non-inferiority analysis, the study demonstrated that the odds ratio (OR) between the two groups was 0.8 (95% CI: 0.4-1.95), indicating no significant difference. Further details are provided in the study's discussion section; p = 0.660, Chi-squared — The p-value was not adjusted for multiple comparisons as there were no multiple outcome measures being compared in this analysis. The significance threshold (alpha) was set at 0.05; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.95], Standard Deviation 18.125 — The standard deviations (SD) for the groups are as follows: For the group receiving 3g fosfomycin: 19.08 For the group receiving 500mg levofloxacin: 17.17; A chi-square test was performed to compare the incidence of UTIs between the two groups: patients receiving a single dose of 500 mg levofloxacin and those receiving a single dose of 3 g fosfomycin, both administered one hour before the urodynamic study (UDS). The result showed no statistically significant difference between the two groups (p = 0.660). An odds ratio was also calculated (OR = 0.8, 95% CI: 0.4-1.95), indicating a slightly lower likelihood of UTI in the fosfomycin group, but the difference was not significant

ADVERSE EVENTS:
Time Frame: After four days of Single Dose Fosfomycin and Single Dose Levofloxacin administration, patients were being assessed for their clinical conditions, such as symptoms related to UTIs, and also adverse events related to Levofloxacin, Fosfomycin administration, and UDS
Description: The adverse events were collected through direct interviews with the patients four days after the procedure.
Arm/Group | Pre-urodynamic Fosfomycin | Pre-urodynamic Levofloxacin
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 3/63 | 2/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-urodynamic Fosfomycin (N=63) | Pre-urodynamic Levofloxacin (N=63)
Nauseous (Gastrointestinal disorders) | 3 (3) | 2 (2) — Five patients reported that they experience nausea after consuming the antibiotics prescribed

LIMITATIONS AND CAVEATS:
The limitation of the study is that many of the patients with UTIs refuse to undergo urine culture tests due to several reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT06017479/Prot_SAP_000.pdf